CLINICAL TRIAL: NCT06197607
Title: Effect of Hand Exercises With and Without Sensory Stimulation on Hand Grip Strength and Manual Ability in Children With Visual Impairment
Brief Title: Effect of Hand Exercises on Hand Grip Strength and Manual Ability in Children With Visual Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/23/0740
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Visual Impairment
Keywords: Hand grip strength; Sensory stimulation; Visual impairment
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Intervention Model Description: Randomised control trial will be conducted with sample size 20. 20 participants will be included in the study. There will be 10 individuals who will receive hand exercises along with sensory stimulation to improve hand grip strength and manual ability and 10 Individuals who will only receive hand exercises to improve hand grip strength and manual ability. Grip strength and will be analyzed using hand dynamometer. For manual dexterity, box and block test will be used. Grip strength and manual dexterity will be analyzed before and after the intervention.Group A individuals will only receive hand exercises to improve hand grip strength and manual ability. Group B individuals will receive hand exercises along with sensory stimulation to improve hand grip strength and manual ability.
Who Masked: Participant
Masking Description: participants will get separate treatment protocols and possible effort will be put to mask the both groups about their treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): The control group will receive thera putty hand exercises.
  Interventions: Other: theraputty hand exercises
- experimental group (Active Comparator): The experimental group will receive sensory stimulation along with theraputty hand exercises.
  Interventions: Other: theraputty hand exercises; Other: sensory stimulation

INTERVENTIONS:
Other: theraputty hand exercises — Theraputty hand exercises will be done in following manners: Finger flexion, Metacarpophalangeal joint flexion, Interphalangeal joint flexion, Finger grip strengthening, Finger abduction and Rolling putty into ball and pinching it between, thumbs and finger with both the hands. There will be 20 repetitions with one set of each
Other: sensory stimulation — Sensory Stimulations (30 min) will be given following forms; All and single joint shaking, Multivariate sensory stimulations, Skin stretch in the muscular region, Fast stretch of the upper limb joints in different directions of motor action, brushing on the large muscles of arm and forearm, brushing on the fingers, Circular massage of the thenar and hypothenar area and pressing the tip of fingers.
  Arms: experimental group

SUMMARY:
Development of the visual system immediately starts after birth via visual stimuli and interactions with the environment. The World Health Organization (WHO) has categorized visual impairments with respect to the best-corrected visual acuity as follows: blindness (Snellen visual acuity of 3/30), severe visual impairment (Snellen visual acuity between 6/60 and 3/30), moderate visual impairment (Snellen visual acuity between 6/18 and 6/60), and mild or no visual impairment (Snellen visual acuity of 6/18). The proper function of hands, particularly in delicate activities, depends on the interaction between the various regions of the brain, particularly, the sensory and motor cortex. Sensory stimulation can be used in such children to improve their manual dexterity and therapeutic interventions can be applied to gain hand strength. Developing skillful hands is a necessity in blind children as it often compensates for their missing vision. This study will focus on effectiveness of hand grip strength and manual ability with sensory stimulation in children with moderate to severe visual impairment.

Theraputty hand exercises and sensory stimulation techniques will be used.

DETAILED DESCRIPTION:
Randomised control trial will be conducted with sample size 20. 20 participants will be included in the study. There will be 10 individuals who will receive hand exercises along with sensory stimulation to improve hand grip strength and manual ability and 10 Individuals who will only receive hand exercises to improve hand grip strength and manual ability. Grip strength and will be analyzed using hand dynamometer. For manual dexterity, box and block test will be used. Grip strength and manual dexterity will be analyzed before and after the intervention.Group A individuals will only receive hand exercises to improve hand grip strength and manual ability. Group B individuals will receive hand exercises along with sensory stimulation to improve hand grip strength and manual ability.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with moderate (Snellen visual acuity between 6/18 and 6/60) to severe (Snellen visual acuity between 6/60 and 3/30) congenital visual impairment. (9)
* Children diagnosed with bilateral congenital visual impairment. (9)
* No prior exposure to therapeutic interventions given to hands. (9)
* Children who can understand English or regional Urdu language. (9)
* Children aged above 6-12 years (9)
* Children of either gender will be included.

Exclusion Criteria:

* Children with any orthopedic problem related to hand. (9)
* Children who went through any surgery of hands or eyes. (9)
* Children with any neurological issues related to hand. (9)
* Those who were unable to communicate or unable to hear well .(5).
* Children diagnosed with complete blindness (Snellen visual acuity of 3/30) .(5).
* Non-co-operative patients

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Box and Block Test (BBT) | 12 weeks
  A rectangular box divided into 2 compartments by a wooden partition is in front of the individual, and 150 coloured wooden blocks are placed in one compartment. The individual is instructed to move as many blocks as possible, one at a time, from one compartment to the other for the duration of 60 seconds. Approximately 5 minutes are required for set up, explanation of the instructions to the patient and administration of the test.
  Stopwatch,Wooden box with partition (box: 53.7 x 25.4 x 8.5 cm, partition: 25.4 cm x 15.2 cm x 1 cm), 150 wooden blocks (2.5 cm cubed).
  Scored by counting the number of blocks carried over by the individual from one compartment to the other. If the individual carries multiple blocks over at a time, this only counts as 1 point.If the individual brings the block over the partition and drops it outside of the box, the block still counts.
Hand Dynamometer | 12 weeks
  : most widely reported device used to measure grip strength. It displays grip force in both pounds and kilograms, with a maximum of 200 lb (90 kg). Handheld dynamometer can ensure quantified strength measurement and clinically, it is very effective and efficient tool. It is also considered as a reliable and valid tool to measure the strength of muscles in the upper and lower extremities. intra-rater (ICC 2, k = 0.95 to 0.97) and inter-rater (ICC 2, k = 0.94 to 0.95) reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Areej Aslam, Ms, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shaikh S. Effect of hand exercises on grip strength and manual dexterity in children with severe congenital visual impairment. Indian Journal of Child Health. 2020;7:477-9